CLINICAL TRIAL: NCT02755012
Title: Reducing Maternal Stress Due to Infection, Malnutrition and Psychosocial Conditions of Poverty: A New Paradigm for Tackling Infant Stunting
Brief Title: Impact of Maternal Stress on Infant Stunting
Status: Completed | Type: Observational
Sponsor: McGill University (Other)
Collaborators: Center for Studies of Sensory Impairment, Aging and Metabolism (Other)
Responsible Party: Principal Investigator, Anne Marie Chomat, Postdoctoral Fellow, McGill University
Other Study IDs: A04-B01-12A
Record Dates: First submitted 2016-04-19; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Maternal; Malnutrition; Infant Malnutrition; Physiological Stress; Emotional Stress; Life Stress; Domestic Violence; Infection; Breast Feeding; Mastitis
Keywords: Maternal Health; Guatemala; Indigenous Population; Stunting; Food Insecurity; Poverty; Social Support; Maternal Autonomy; Paternal Support; Cortisol Rhythm
MeSH Terms: conditions — Malnutrition; Infant Nutrition Disorders; Stress, Psychological; Infections; Breast Feeding; Mastitis; Growth Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool sample (mother and infant) Urine sample (mother) Saliva sample (mother) Breast milk sample (mother)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Longitudinal: 155 women enrolled in 2nd or 3rd trimester of pregnancy, and seen again, with their infant, at 0-6 wk postpartum, and 4-6 mo postpartum
- Early Postpartum: 60 women enrolled at 0-6 wk postpartum and seen once with their infant (cross-sectional)
- Later Postpartum: 56 women enrolled at 0-6 wk postpartum and seen once with their infant (cross-sectional)

SUMMARY:
This study takes place in rural Mam-Mayan communities of Guatemala characterized by high rates of childhood stunting. It aims to characterize women's exposure to nutrition, infection and psychosocial stressors vs. resilience factors, to evaluate the cumulative impact of maternal-level factors (nutritional, infectious, psychosocial), social factors (autonomy, social support, domestic violence), and household factors (socioeconomic status, food security) on early infant growth, and to evaluate whether maternal cortisol may be a mediator in the vertical transmission of stress.

DETAILED DESCRIPTION:
Grounded in participatory action research and a socio-ecological framework, this mixed-methods, observational study enrolled a longitudinal cohort of 155 women, seen during pregnancy (6-9 mo), early (0-6 wks) and later (4-6 mo) postpartum, and two cross-sectional cohorts (60 early, 56 later postpartum).

Maternal and infant anthropometry was recorded, maternal fecal, urine and saliva samples were collected, and questionnaires were used to explore household factors (socioeconomic status, food security), social factors (autonomy, paternal/social support, domestic violence), and maternal-level factors (nutrition, infection, emotional distress).

Analyses focused on (1) characterizing women's exposure to nutrition, infection and psychosocial stressors vs. resilience factors, (2) describing the maternal diurnal salivary cortisol rhythm in pregnancy and postpartum and explore its association with psychosocial variables, (3) assessing the cumulative impact of maternal-level factors (nutritional, infectious, psychosocial), social factors (autonomy, social support, domestic violence), and household factors (socioeconomic status, food security) on early infant growth, and (4) evaluating whether maternal cortisol may be a mediator in the vertical transmission of stress.

In addition, Photovoice activities involved giving a camera to 23 women from study communities, who documented sources of stress vs. resilience for local women, and shared photo-elicited narratives through six group sessions.

ELIGIBILITY:
Inclusion Criteria:

* Woman from study communities
* Either pregnant or 0-6 wk postpartum or 4-6 mo postpartum
* Consenting to participate

Exclusion Criteria:

* Twin pregnancy
* Not consenting to participate

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Indigenous Mam-Mayan women living in 8 rural hamlets (or communities) in the municipality of San Juan Ostuncalco, in the department of Quetzaltenango, Guatemala.
Sampling Method: Non-Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Infant stunting (Infant height-for-age score) | 0-6 wk
  Infant height-for-age score measured at 0-6 wk
Infant stunting (Infant height-for-age score) | 4-6 mo postpartum
  Infant height-for-age score measured at 4-6 mo postpartum
Change in infant HAZ per month | Change over time (between 0-6wk and 4-6mo)
  Change in infant HAZ score between 1st (0-6 wk) and 2nd (4-6 mo) visits

CONTACTS AND LOCATIONS:
Overall Officials: Anne Marie Chomat, MD, PhD, MPH, Principal Investigator — McGill University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chomat AM, Solomons NW, Koski KG, Wren HM, Vossenaar M, Scott ME. Quantitative Methodologies Reveal a Diversity of Nutrition, Infection/Illness, and Psychosocial Stressors During Pregnancy and Lactation in Rural Mam-Mayan Mother-Infant Dyads From the Western Highlands of Guatemala. Food Nutr Bull. 2015 Dec;36(4):415-40. doi: 10.1177/0379572115610944. Epub 2015 Oct 19. PMID 26481796
- [Result] Solomons NW, Vossenaar M, Chomat AM, Doak CM, Koski KG, Scott ME. Stunting at birth: recognition of early-life linear growth failure in the western highlands of Guatemala. Public Health Nutr. 2015 Jul;18(10):1737-45. doi: 10.1017/S136898001400264X. PMID 26017476
- [Result] Wren HM, Solomons NW, Chomat AM, Scott ME, Koski KG. Cultural determinants of optimal breastfeeding practices among indigenous Mam-Mayan women in the Western Highlands of Guatemala. J Hum Lact. 2015 Feb;31(1):172-84. doi: 10.1177/0890334414560194. PMID 25583316